CLINICAL TRIAL: NCT06759558
Title: Allopregnanolone (Zuranolone) in Post-stroke Depression
Acronym: ALLO in PSD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00118406
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Post Stroke Depression
Keywords: zuranolone; post stroke depression; allopregnanolone; stroke
MeSH Terms: conditions — Stroke | interventions — zuranolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Zuranolone (Experimental): Participants in the Zuranolone arm will be treated for post-stroke depression for 14 days with 50mg of zuranolone once daily.
  Interventions: Drug: Zuranolone

INTERVENTIONS:
Drug: Zuranolone — Zuranolone is a neuroactive steroid that works by modulating the activity of the gamma-aminobutyric acid (GABA) receptor in the brain.

SUMMARY:
The goal of this Phase II clinical trial is to learn if the oral synthetic allopreganolone analog (zuranolone) is safe to take and is well tolerated by stroke survivors experiencing moderate to severe post-stroke depression and if it will help with the symptoms of depression. The main questions it will aim to answer are:

* Is zuranolone safe to take by participants who have moderate to severe post-stroke depression?
* Is zuranolone well-tolerated by participants who have moderate to severe post-stroke depression?
* Does zuranolone treat moderate to severe post-stroke depression?

The study will enroll six participants. All participants will be given 50 mg of zuranolone for 14 days.

Participants will be asked to provide blood samples, complete some questionnaires including those related to mood and a cognitive assessment.

ELIGIBILITY:
Inclusion Criteria:

* 21-65 years old of any sex and race/ethnicity
* Clinical ischemic or hemorrhagic acute stroke (confirmed by CT or MRI) occurring within 1 year of date of enrollment
* Moderate to severe PSD (Post-Stroke Depression) defined as having depressive symptoms lasting for at least 2 weeks and scoring 17 or more on the HAM-D (Hamilton Depression Rating Scale)

Exclusion Criteria:

* Have abused or been dependent on narcotics, recreational drug use, or alcohol
* Advanced liver or kidney problems
* Pregnant or plan to become pregnant
* Post-partum period or breastfeeding
* History of attempted suicide
* Active psychosis or suicidal ideation necessitating clinical intervention
* Antidepressant medications titration or initiation within 12 weeks of recruitment
* History of Bipolar disorder, schizophrenia or treatment resistant depression preceding the stroke

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-01-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events (TEAEs) after starting zuranolone | 90 days
  TEAEs: suicidality and signs of abuse/dependence such as suicidal thinking and associated behaviors, such as anxiety, agitation, panic attacks, insomnia, irritability, hostility, impulsivity, akathisia, hypomania, and mania, psychosis, worsening depression.
  Other TEAEs include: dizziness, somnolence, significant drowsiness causing impairment of daily activity, skin rash, abdominal pain, diarrhea, urinary tract infection, fatigue, memory impairment, tremor, muscle twitching, myalgia, headache, hypoesthesia, recurrent stroke, hypertension, hypotension, falls, confusion.
Severity of suicidal ideation after starting zuranolone as measured by the Columbia Suicide Severity Rating Scale (C-SSRS) | 90 Days
  The C-SSRS will be used to evaluate the intensity of suicidal ideation. The score ranges from 2 to 25, where a higher score indicates greater ideation.
Severity of somnolence after starting zuranolone as measured by the Epworth Sleepiness Scale (ESS) | 90 Days
  The ESS will be used to evaluate the intensity of somnolence. The score ranges from 0 to 24, where a score from 11-24 indicates excessive daytime sleepiness.

SECONDARY OUTCOMES:
Change from baseline in Hamilton Depression Rating Scale (HAM-D) score at days 15 and 90 | Baseline, 15 days, 90 days
  A mixed-effects model for repeated measures will be used for the secondary exploratory outcome and will include change from baseline in HAM-D at each visit as the dependent variable. Logistic regression models for repeated measures using the generalized estimating equation method will be applied for analysis of HAM-D response and HAM-D remission.
  HAM-D score ranges from 0-50. In general the higher the total score the more severe the depression.
Change from baseline in Hamilton Anxiety Rating Scale (HAM-A) score at days 15 and 90 | Baseline, 15 days, 90 days
  The HAM-A total score ranges from 0 to 56, with higher scores indicating greater anxiety.
Number of participants with HAM-D response at 3, 15, and 90 days | 3 days, 15 days, 90 days
  The HAM-D total score ranges from 0 to 54, with higher scores indicating greater severity of depression. Response is defined as having a > or = 50% score reduction.
Number of participants with HAM-D remission (score ≤7) rates at 3, 15, and 90 days | 3 days, 15 days, 90 days
  The HAM-D total score ranges from 0 to 54, with higher scores indicating greater severity of depression. Remission is defined as having a score < or = 7.

CONTACTS AND LOCATIONS:
Overall Officials: Nada El Husseini, MD, Principal Investigator — Duke University
Locations (1):
- Duke South Neurology Clinic 1L, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared via publications and/or presentations

REFERENCES:
- [Background] Wang S, Zhang W, Liu Z, Zhang T, Wang Y, Li W. Efficacy and safety of zuranolone in the treatment of major depressive disorder: a meta-analysis. Front Neurosci. 2024 Jan 16;17:1332329. doi: 10.3389/fnins.2023.1332329. eCollection 2023. PMID 38292895
- [Background] Clayton AH, Lasser R, Parikh SV, Iosifescu DV, Jung J, Kotecha M, Forrestal F, Jonas J, Kanes SJ, Doherty J. Zuranolone for the Treatment of Adults With Major Depressive Disorder: A Randomized, Placebo-Controlled Phase 3 Trial. Am J Psychiatry. 2023 Sep 1;180(9):676-684. doi: 10.1176/appi.ajp.20220459. Epub 2023 May 3. PMID 37132201
- [Background] Deligiannidis KM, Meltzer-Brody S, Gunduz-Bruce H, Doherty J, Jonas J, Li S, Sankoh AJ, Silber C, Campbell AD, Werneburg B, Kanes SJ, Lasser R. Effect of Zuranolone vs Placebo in Postpartum Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2021 Sep 1;78(9):951-959. doi: 10.1001/jamapsychiatry.2021.1559. PMID 34190962
- [Background] Sripada RK, Marx CE, King AP, Rampton JC, Ho SS, Liberzon I. Allopregnanolone elevations following pregnenolone administration are associated with enhanced activation of emotion regulation neurocircuits. Biol Psychiatry. 2013 Jun 1;73(11):1045-53. doi: 10.1016/j.biopsych.2012.12.008. Epub 2013 Jan 21. PMID 23348009
- [Background] Chen S, Gao L, Li X, Ye Y. Allopregnanolone in mood disorders: Mechanism and therapeutic development. Pharmacol Res. 2021 Jul;169:105682. doi: 10.1016/j.phrs.2021.105682. Epub 2021 May 18. PMID 34019980
- [Background] Pinna G, Almeida FB, Davis JM. Allopregnanolone in Postpartum Depression. Front Glob Womens Health. 2022 Apr 26;3:823616. doi: 10.3389/fgwh.2022.823616. eCollection 2022. PMID 35558166
- [Background] Diviccaro S, Cioffi L, Falvo E, Giatti S, Melcangi RC. Allopregnanolone: An overview on its synthesis and effects. J Neuroendocrinol. 2022 Feb;34(2):e12996. doi: 10.1111/jne.12996. Epub 2021 Jun 29. PMID 34189791
- [Background] Chen S, Wang T, Yao J, Brinton RD. Allopregnanolone Promotes Neuronal and Oligodendrocyte Differentiation In Vitro and In Vivo: Therapeutic Implication for Alzheimer's Disease. Neurotherapeutics. 2020 Oct;17(4):1813-1824. doi: 10.1007/s13311-020-00874-x. PMID 32632771
- [Background] Dymm B, Goldstein LB, Unnithan S, Al-Khalidi HR, Koltai D, Bushnell C, Husseini NE. Depression following small vessel stroke is common and more prevalent in women. J Stroke Cerebrovasc Dis. 2024 May;33(5):107646. doi: 10.1016/j.jstrokecerebrovasdis.2024.107646. Epub 2024 Feb 22. PMID 38395097
- [Background] El Husseini N, Goldstein LB, Peterson ED, Zhao X, Olson DM, Williams JW Jr, Bushnell C, Laskowitz DT. Depression Status Is Associated with Functional Decline Over 1-Year Following Acute Stroke. J Stroke Cerebrovasc Dis. 2017 Jul;26(7):1393-1399. doi: 10.1016/j.jstrokecerebrovasdis.2017.03.026. Epub 2017 Apr 25. PMID 28389192
- [Background] Redmond C, Bushnell C, Duncan P, D'Agostino R Jr, Ambrosius WT, Bishop L, Gesell S, Prvu-Bettger J, El Husseini N. Association of in-hospital depression and anxiety symptoms following stroke with 3 months- depression, anxiety and functional outcome. J Clin Neurosci. 2022 Apr;98:133-136. doi: 10.1016/j.jocn.2022.02.010. Epub 2022 Feb 15. PMID 35180502
- [Background] El Husseini N, Goldstein LB, Peterson ED, Zhao X, Pan W, Olson DM, Zimmer LO, Williams JW Jr, Bushnell C, Laskowitz DT. Depression and antidepressant use after stroke and transient ischemic attack. Stroke. 2012 Jun;43(6):1609-16. doi: 10.1161/STROKEAHA.111.643130. Epub 2012 Mar 29. PMID 22461330
- [Background] Schottke H, Giabbiconi CM. Post-stroke depression and post-stroke anxiety: prevalence and predictors. Int Psychogeriatr. 2015 Nov;27(11):1805-12. doi: 10.1017/S1041610215000988. Epub 2015 Jul 16. PMID 26178418
- [Background] Xu J, Zhou Y, Yan C, Wang X, Lou J, Luo Y, Gao S, Wang J, Wu L, Gao X, Shao A. Neurosteroids: A novel promise for the treatment of stroke and post-stroke complications. J Neurochem. 2022 Jan;160(1):113-127. doi: 10.1111/jnc.15503. Epub 2021 Sep 21. PMID 34482541
- [Background] Ishrat T, Sayeed I, Atif F, Hua F, Stein DG. Progesterone and allopregnanolone attenuate blood-brain barrier dysfunction following permanent focal ischemia by regulating the expression of matrix metalloproteinases. Exp Neurol. 2010 Nov;226(1):183-90. doi: 10.1016/j.expneurol.2010.08.023. Epub 2010 Sep 15. PMID 20816826
- [Background] Rauch SAM, Sripada R, Burton M, Michopoulos V, Kerley K, Marx CE, Kilts JD, Naylor JC, Rothbaum BO, McLean CP, Smith A, Norrholm SD, Jovanovic T, Liberzon I, Williamson DE, Yarvis CJS, Dondanville KA, Young-McCaughan S, Keane TM, Peterson AL; Consortium to Alleviate PTSD and the STRONG STAR Consortium. Neuroendocrine biomarkers of prolonged exposure treatment response in military-related PTSD. Psychoneuroendocrinology. 2020 Sep;119:104749. doi: 10.1016/j.psyneuen.2020.104749. Epub 2020 Jun 8. PMID 32554173
- [Background] Kinzel P, Marx CE, Sollmann N, Hartl E, Guenette JP, Kaufmann D, Bouix S, Pasternak O, Rathi Y, Coleman MJ, van der Kouwe A, Helmer K, Kilts JD, Naylor JC, Morey RA, Shutter L, Andaluz N, Coimbra R, Lang AJ, George MS, McAllister TW, Zafonte R, Stein MB, Shenton ME, Koerte IK. Serum Neurosteroid Levels Are Associated With Cortical Thickness in Individuals Diagnosed With Posttraumatic Stress Disorder and History of Mild Traumatic Brain Injury. Clin EEG Neurosci. 2020 Jul;51(4):285-299. doi: 10.1177/1550059420909676. Epub 2020 Mar 18. PMID 32186207
- [Background] Umminger LF, Rojczyk P, Seitz-Holland J, Sollmann N, Kaufmann E, Kinzel P, Zhang F, Kochsiek J, Langhein M, Kim CL, Wiegand TLT, Kilts JD, Naylor JC, Grant GA, Rathi Y, Coleman MJ, Bouix S, Tripodis Y, Pasternak O, George MS, McAllister TW, Zafonte R, Stein MB, O'Donnell LJ, Marx CE, Shenton ME, Koerte IK. White Matter Microstructure Is Associated with Serum Neuroactive Steroids and Psychological Functioning. J Neurotrauma. 2023 Apr;40(7-8):649-664. doi: 10.1089/neu.2022.0111. Epub 2023 Jan 6. PMID 36324218
- [Background] Pibiri F, Nelson M, Guidotti A, Costa E, Pinna G. Decreased corticolimbic allopregnanolone expression during social isolation enhances contextual fear: A model relevant for posttraumatic stress disorder. Proc Natl Acad Sci U S A. 2008 Apr 8;105(14):5567-72. doi: 10.1073/pnas.0801853105. Epub 2008 Apr 7. PMID 18391192
- [Background] Pisu MG, Garau A, Olla P, Biggio F, Utzeri C, Dore R, Serra M. Altered stress responsiveness and hypothalamic-pituitary-adrenal axis function in male rat offspring of socially isolated parents. J Neurochem. 2013 Aug;126(4):493-502. doi: 10.1111/jnc.12273. Epub 2013 May 9. PMID 23600845
- [Background] Almeida FB, Nin MS, Barros HMT. The role of allopregnanolone in depressive-like behaviors: Focus on neurotrophic proteins. Neurobiol Stress. 2020 Apr 9;12:100218. doi: 10.1016/j.ynstr.2020.100218. eCollection 2020 May. PMID 32435667
- [Background] Hellgren C, Akerud H, Skalkidou A, Backstrom T, Sundstrom-Poromaa I. Low serum allopregnanolone is associated with symptoms of depression in late pregnancy. Neuropsychobiology. 2014;69(3):147-53. doi: 10.1159/000358838. Epub 2014 Apr 26. PMID 24776841
- [Background] Osborne LM, Gispen F, Sanyal A, Yenokyan G, Meilman S, Payne JL. Lower allopregnanolone during pregnancy predicts postpartum depression: An exploratory study. Psychoneuroendocrinology. 2017 May;79:116-121. doi: 10.1016/j.psyneuen.2017.02.012. Epub 2017 Feb 16. PMID 28278440
- [Background] He J, Evans CO, Hoffman SW, Oyesiku NM, Stein DG. Progesterone and allopregnanolone reduce inflammatory cytokines after traumatic brain injury. Exp Neurol. 2004 Oct;189(2):404-12. doi: 10.1016/j.expneurol.2004.06.008. PMID 15380490
- [Background] Xilouri M, Papazafiri P. Anti-apoptotic effects of allopregnanolone on P19 neurons. Eur J Neurosci. 2006 Jan;23(1):43-54. doi: 10.1111/j.1460-9568.2005.04548.x. PMID 16420414
- [Background] Paul SM, Pinna G, Guidotti A. Allopregnanolone: From molecular pathophysiology to therapeutics. A historical perspective. Neurobiol Stress. 2020 Mar 14;12:100215. doi: 10.1016/j.ynstr.2020.100215. eCollection 2020 May. PMID 32435665
- [Background] Schule C, Nothdurfter C, Rupprecht R. The role of allopregnanolone in depression and anxiety. Prog Neurobiol. 2014 Feb;113:79-87. doi: 10.1016/j.pneurobio.2013.09.003. Epub 2013 Nov 8. PMID 24215796
- [Background] Wang M. Neurosteroids and GABA-A Receptor Function. Front Endocrinol (Lausanne). 2011 Oct 4;2:44. doi: 10.3389/fendo.2011.00044. eCollection 2011. PMID 22654809
- [Background] El Husseini N, Laskowitz DT. The role of neuroendocrine pathways in prognosis after stroke. Expert Rev Neurother. 2014 Feb;14(2):217-32. doi: 10.1586/14737175.2014.877841. Epub 2014 Jan 13. PMID 24428141
- [Background] Towfighi A, Ovbiagele B, El Husseini N, Hackett ML, Jorge RE, Kissela BM, Mitchell PH, Skolarus LE, Whooley MA, Williams LS; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; and Council on Quality of Care and Outcomes Research. Poststroke Depression: A Scientific Statement for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2017 Feb;48(2):e30-e43. doi: 10.1161/STR.0000000000000113. Epub 2016 Dec 8. PMID 27932603